CLINICAL TRIAL: NCT02998047
Title: A Phase I Study of Lintuzumab-Ac225 in Patients With Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Actinium Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lin-AC225-MM01
Record Dates: First submitted 2016-12-12; First posted 2016-12-20 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IV infusion of Lintuzumab AC225 (Experimental): Starting dose - 0.5 μCi/Kg IV infusion of Lintuzumab AC225 on Day 1 of each cycle with dose escalation 1 μCi/Kg and 1.5 μCi/Kg or de-escalation to 0.25 μCi/Kg.
  1 cycle = 28 days, up to 3 to 8 cycles (depending on the cohort).
  Interventions: Drug: Lintuzumab AC 225

INTERVENTIONS:
Drug: Lintuzumab AC 225 — Lintuzumab-Ac225 is an immunoconjugate [antibody: anti-CD 33 antibody and radioactive isotope: Actinium (225Ac)] for the treatment of multiple myeloma.
  Other Names: HuM195-Ac225

SUMMARY:
1. Establish the MTD of Lintuzumab-Ac225 as monotherapy
2. Establish overall response rate (ORR) where ORR = CR + sCR+ VGPR+PR)
3. Confirm the safety profile of the treatment regimen
4. Estimate progression-free survival (PFS) and overall survival

DETAILED DESCRIPTION:
The study is a multicenter, open label Phase I trial. Phase 1, dose-escalation : This study uses a 3+3 design to estimate the maximum tolerated dose (MTD).

There will be 3 escalating dose levels in the trial (0.5 μCi/kg, 1 μCi/kg, and 1.5 μCi/kg). Each dose can be administered in up to 3-8 cycles providing that the total dose received per patient does not exceed 4.5 μCi/kg.

De-escalation (decrease dose level to 0.25 μCi/kg) is planned if at the first dose level of 0.5 μCi/kg, after expanding the cohort to a maximum of 6 patients, ≥2 patient have DLTs. At the dose level of 0.25 μCi/kg, if eligible to continue receiving additional doses of the study drug, patients will receive up to 8 doses in total, with the total administered activity being 2 μCi/kg.

The starting dose level will be 0.5 μCi/kg of 225Ac-Lintuzumab administered on day 1 of each cycle. If this dose level is safe, the second dose level of 1 μCi/kg will be explored. If the starting dose level results in DLTs in ≥2 patients, the dose level of 0.25 μCi/kg will be explored.

Subjects will receive the investigational drug as a single infusion at the prescribed dose level.

Intra cohort dose escalation/ decrease is not allowed.

Minimum three to maximum six patients will be treated at each dose level, and dose escalation will proceed as follows:

1. Rules for dose escalation are:

   1. If 0 of 3 patients have a DLT, escalate to the next dose level (Unless enrolling patients at the 0.25 µCi/kg dose level)
   2. If 1 of 3 patients has a DLT, expand the cohort to 6 patients
   3. If ≤1 of 6 patients has a DLT, escalate to the next dose level (Unless enrolling patients at the 0.25 µCi/kg dose level)
   4. If ≥2 of 3 or ≥2 of 6 patients have a DLT, then the previous dose is the MTD (Unless enrolling patients at the 0.25 µCi/kg level, in which case the trial is terminated)
   5. Three patients will start at the 0.50 uCi/kg dose. The next dose level will be 1.0 µCi/kg and the final dose level will be 1.5 µCi/kg. Dose de-escalation to 0.25 µCi/kg will occur if, at the 0.5 µCi/kg dose, there are ≥2 of 3 or ≥2 of 6 patients with a DLT.
2. If a patient has not progressed nor had CR by the end of a cycle, the patient can continue treatment for a maximum of three (1.5 µCi/kg), four (1.0 µCi/kg), or eight cycles (0.25 µCi/kg and 0.50 µCi/kg).

All patients may receive GCSF support starting on Day 9 if clinically indicated and continuing until ANC>1,000.

After the dose escalation portion is completed, treat 3 additional patients at the highest established dose level to confirm MTD and establish that dose level as MTD.

ELIGIBILITY:
Inclusion Criteria-

* Confirmed diagnosis of multiple myeloma with measurable disease, as defined by the presence of M immunoglobulin protein in serum electrophoresis of at least 0.5 g/dL for IgG or 0.5 g/dL for IgA or urinary excretion of at least 200 mg monoclonal light chain per 24 hours.
* Clinical diagnosis of multiple myeloma requiring treatment that has relapsed after or proven refractory to at least three prior treatment regimens, and in the opinion of the investigator must not be candidates for any FDA approved drug known to provide clinical benefit.
* All acute toxicities from any prior therapy (radiotherapy, chemotherapy, or surgical procedures) resolved to Grade ≤ 2, NCI CTCAE.
* Serum potassium and magnesium levels within institutional normal limits. Total serum calcium or ionized calcium level must be greater than or equal to the lower limit of normal.
* Greater than 25% of myeloma plasmocytes from bone marrow must be CD33 positive.
* Required baseline laboratory data including: White blood cell count, Absolute neutrophil count (ANC), Platelets, Hemoglobin, Serum creatinine, AST, Creatinine clearance, Bilirubin , AST and ALT , FEV1/FVC
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2

Exclusion Criteria-

* Sex and Reproductive Status

  * Women of child bearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least one month (4 weeks) before and for at least six months (6 months) after the last dose of study medication.
  * Women who are pregnant or breastfeeding
  * Women with a positive pregnancy test on enrollment or prior to investigational product administration.
  * Men whose sexual partners are WOCBP, who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least six months (6 months) after completion of study medication.
* Target Disease Exceptions

  * Concurrent therapy with any other investigational agent.
  * Concomitant therapy with bisphosphonates.
  * Pathological fracture within 3 months prior to treatment;
  * Symptomatic spinal cord compression; .
* Medical History and Concurrent Diseases

  * Treatment with chemotherapy or biological therapy 3 weeks prior to enrollment;
  * Presence of HAHA on screening
  * No bone marrow transplant within 3 months prior to treatment initiation
  * Prior treatment with radiation to cumulative maximum tolerated dose
  * Clinically significant cardiac disease (NYHA Class III or IV) including preexisting arrhythmia (such as ventricular tachycardia, ventricular fibrillation, or "Torsade de Pointes")
  * Myocardial infarction, uncontrolled angina within 6 months, congestive heart failure, or cardiomyopathy.
  * Abnormal QTc interval prolonged (> 450 msec) after electrolytes have been corrected on baseline ECG.
  * Clinically significant pleural effusion in the previous 12 months or current ascites.
  * Clinically-significant coagulation or platelet function disorder (eg, known von Willebrand's disease).
  * Prior or concurrent malignancy, except for the following:

    i) Adequately treated basal cell or squamous cell skin cancer ii) Cervical carcinoma in situ iii) Adequately treated Stage I or II cancer from which the subject is currently in complete remission iv) Or any other cancer from which the subject has been disease-free for 3 years.
* Physical and Laboratory Test Findings

  o Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality, serious uncontrolled medical disorder or active infection that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for this study.
* Allergies and Adverse Drug Reactions

  o Intolerance to humanized monoclonal antibodies
* Other Exclusion Criteria

  * Prisoners or subjects who are involuntarily incarcerated.
  * Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
* Treatment with radiation within 6 weeks
* Active serious infections uncontrolled by antibiotics
* Clinically significant pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-12; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated dose of Lintuzumab-AC225 | Through study completion, an average of 2.5 year
  establish the maximum tolerated dose as monotherapy
Adverse events- Treatment Emergent | Through study completion, an average of 2.5 year
  safety of lintuzumab-Ac225

SECONDARY OUTCOMES:
Response rates (objective response rate, complete response rate, stringent complete response rate, very good partial response rate and partial response rate) | Through study completion, an average of 2.5 year
  response rate, including ORR, CR, sCR, VGPR, and PR, PFS, and OS. Efficacy assessments will include serum and urine analyses for paraprotein levels and bone marrow analyses.
Progression free survival | Through study completion, an average of 2.5 year
  Progression free survival
Overall survival | Through study completion, an average of 2.5 year
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Avinash Desai, MD, Study Director — Actinium Pharmaceuticals
Locations (5):
- United States (5):
  - UCLA, Los Angeles, California
  - University Of Kansas Medical Center, Kansas City, Kansas
  - Memorial Sloan Kettering Cancer CEnter, New York, New York
  - Baylor Scott and White Research Institute, Charles A. Sammons Cancer Center, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No